CLINICAL TRIAL: NCT02457078
Title: Investigating the Effects of Nutrition on the Maturation of Brain Networks Associated With Memory and Language in Infants
Brief Title: Investigating the Effects of Nutrition on the Maturation of Brain Networks Associated With Memory in Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANGC1401
Record Dates: First submitted 2015-02-05; First posted 2015-05-29 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Healthy
Keywords: nutritional supplements; lutein; DHA; vitamin E; infant brain development

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Postnatal Dietary Supplement (Experimental): Dietary Supplement: docosahexaenoic acid, lutein, and α-tocopherol (vitamin E). 1 capsule per day will be consumed beginning immediately after birth and continuing for 9 months.
  Interventions: Dietary Supplement: Postnatal Dietary Supplement
- Control Supplement (Placebo Comparator): Control Supplement: Capsule containing soybean oil and α-tocopheryl (vitamin E). 1 capsule per day will be consumed beginning immediately after birth and continuing for 9 months.
  Interventions: Dietary Supplement: Control Supplement

INTERVENTIONS:
Dietary Supplement: Postnatal Dietary Supplement — Dietary Supplement: docosahexaenoic acid, lutein, and α-tocopherol (vitamin E). 1 capsule per day will be consumed beginning immediately after birth and continuing for 9 months.
  Arms: Postnatal Dietary Supplement
Dietary Supplement: Control Supplement — Placebo Supplement:soybean oil and α-tocopherol (vitamin E)
  Arms: Control Supplement

SUMMARY:
This project will investigate whether adding nutritional supplements to the diet will have beneficial effects on the development of infant brain networks (assessed at 4 and 9 months of age). The nutritional supplement will contain lutein (typically found in leafy vegetables),docosahexaenoic acid (DHA; a fatty acid typically found in cold-water fish such as salmon or tuna), and of vitamin E.

DETAILED DESCRIPTION:
This project will investigate whether adding nutritional supplements to the diet will have beneficial effects on the development of infant brain networks (assessed at 4 and 9 months of age). The nutritional supplement will contain lutein (typically found in leafy vegetables),docosahexaenoic acid (DHA; a fatty acid typically found in cold-water fish such as salmon or tuna), and of vitamin E. This supplement will be taken orally, once a day for 9-10 months starting immediately after delivery. The investigators will also collect a dry blood spot (DBS) from the heel of the infant at 4 and 9 months of age to assess the amount of these nutrients reaching the infants' blood. At these same ages, the investigators will use the Event-Related Optical Signal (EROS) to non-invasively record brain activity in the infants as they passively listen to sounds (e.g., novel sounds, speech sounds, words, etc.) and watch short video clips of moving objects (e.g., toys, children playing, etc) to look at whether the nutritional supplement influences brain development.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for mothers at time of recruitment:

  1. Intention to breast feed for at least the first 3 months
  2. 18 years of age or older
  3. Willingness to abstain from multi-vitamins or other supplements that contain lutein and vitamin E during the study and take no more than 200 mg of DHA.
  4. Normal or corrected-to-normal vision
  5. Normal or corrected-to-normal hearing
  6. English is the dominant language spoken in the home.

Exclusion Criteria:

* and/or early termination:

  1. Mother is taking cholesterol medication and/or medication affecting lipid absorption and/or transport.
  2. High risk pregnant mothers
  3. Macular Pigment Optical Density (MPOD) score greater than 0.6.
  4. Preterm birth (less than 37 weeks)
  5. Low birth weight (less than 2500 grams, < 5.5 pounds)
  6. Unable or unwilling to continue breast feeding within the first 3 months after birth.
  7. Unable or unwilling to continue taking the study supplement within the first 3 months after birth.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Brain Imaging (Event-Related Optical Signal) of breastfed 4 month old infant | Brain activity will be assessed at 4 months of age
  The current project will investigate whether nutritional supplements will have beneficial effects on infant brain networks at 4 months of age. We will use the Event-Related Optical Signal (EROS) to non-invasively record brain activity in the infants as they passively listen to sounds (e.g., novel sounds, speech sounds, words, etc.) and watch short video clips of moving objects (e.g., toys, children playing, etc) to look at whether the nutritional supplement influences brain development.
Brain Imaging (Event-Related Optical Signal) of breastfed 9 month old infant | Brain activity will be assessed at 9 months of age
  The current project will investigate whether nutritional supplements will have beneficial effects on infant brain networks at 9 months of age. We will use the Event-Related Optical Signal (EROS) to non-invasively record brain activity in the infants as they passively listen to sounds (e.g., novel sounds, speech sounds, words, etc.) and watch short video clips of moving objects (e.g., toys, children playing, etc) to look at whether the nutritional supplement influences brain development.

SECONDARY OUTCOMES:
Infant Dry Blood Spot at 4 months | 4 months of age
  We will also collect a dry blood spot (DBS) from the heel of the infant at 4 months of age to assess the amount of the nutrients reaching the infants' blood.
Infant Dry Blood Spot at 9 months | 9 months of age
  We will also collect a dry blood spot (DBS) from the heel of the infant at 9 months of age to assess the amount of the nutrients reaching the infants' blood.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Gratton, Ph.D., M.D., Principal Investigator — University of Illinois at Chicago
Locations (1):
- Beckman Institute, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sherry CL, Oliver JS, Renzi LM, Marriage BJ. Lutein supplementation increases breast milk and plasma lutein concentrations in lactating women and infant plasma concentrations but does not affect other carotenoids. J Nutr. 2014 Aug;144(8):1256-63. doi: 10.3945/jn.114.192914. Epub 2014 Jun 4. PMID 24899160
- [Background] Gratton G, Fabiani M. Fast optical imaging of human brain function. Front Hum Neurosci. 2010 Jun 23;4:52. doi: 10.3389/fnhum.2010.00052. eCollection 2010. PMID 20631845